CLINICAL TRIAL: NCT02790970
Title: Interventional, Randomised, Open Label, Multi-centre, Parallel-group, Controlled Study Investigating the Effects of Using the PReDicT Test to Guide the Antidepressant Treatment of Depressed Patients
Brief Title: Predicting Response to Depression Treatment (PReDicT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: P1vital Products Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P1V-DEP-MD03
Record Dates: First submitted 2016-03-30; First posted 2016-06-06 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PReDicT Test (Experimental): To determine whether use of the PReDicT Test to direct antidepressant treatment results in an increased proportion of depressed patients showing a response to treatment at week 8
  Interventions: Device: PReDicT Test
- Treatment as usual (Placebo Comparator): Treat patients as usual without using the predict test to determine treatment.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Device: PReDicT Test — PReDicT Test, when completed 7-9 days after starting antidepressant treatment, is able to predict a patient's subsequent response to that antidepressant treatment 4-6 weeks later
  Arms: PReDicT Test
Other: Treatment as Usual — Patients treated by the clinician conventionally using signs and symptoms to determine treatment changes or medication changes.
  Arms: Treatment as usual

SUMMARY:
Depression is a very common, serious and in some cases life-threatening condition, affecting around 350 million people globally. Approximately 11% of citizens in the European Union suffer from depression at some point in their lives. Depression is associated with significant socio-economic costs and has been predicted to become the greatest cause of disability worldwide by 2030 . In 2010 it was estimated that there were approximately 30 million patients with depression in Europe, with aggregated economic costs of approximately €92 billion . Improvements in managing the treatment of depression are urgently needed to improve patient outcomes, contain rising healthcare costs, improve workplace productivity and help to address global economic and societal challenges.

While a range of effective antidepressant medications are available to treat depression, it takes 4-6 weeks after starting antidepressant treatment before a physician can detect whether the treatment is working. However, surprisingly, more than 50% of patients fail to respond to the first antidepressant treatment they are prescribed. Therefore, it often takes several months to identify an effective antidepressant treatment for the majority of patients with depression. During this time a patient's ability to work and function socially is severely impaired. Individuals may be absent from work for many weeks or months and this places a substantial burden on the economy and on healthcare resources.

DETAILED DESCRIPTION:
The study is a randomized, two-arm, multi-centre, open label, clinical investigation of a medical device, the Predicting Response to Depression Treatment Test (PReDicT Test) . It will be conducted in depressed patients in primary care settings in five European countries (UK, France, Spain, Germany and the Netherlands).

The study is divided into an 8 to 10 week clinical phase and a 40 week follow-up phase. Each participant will be in the study for a total of up to 48-50 weeks.

During the clinical phase, participants will attend between 2 and 4 study visits, depending on their study arm and their response to treatment. Some of these visits may be conducted by telephone. Participants will also complete weekly online questionnaires from home.

During the follow-up phase participants will complete online questionnaires from home every 4 weeks over a 40 week period. Study visits will not be required during the follow-up phase.

An electronic Patient Reported Outcomes (ePRO) system, accessed via a study website, will be used to collect questionnaire data and PReDicT Test responses. The ePRO system will be used to randomise participants and will issue email reminders to participants and study researchers when study-related activities are due.

Visit 1: Screening and PReDicT #1 The visit will take place at the study site 0 to 7 days after the SSRI was prescribed. Visit 1 may take place on the same day as the Selective Serotonin Reuptake Inhibitor (SSRI) was prescribed only if local approvals permit this to happen. Informed Consent must be obtained before any study procedures are performed. Visit duration will be approximately 90 minutes.

The following will take place at Visit 1:

* Informed Consent
* Unique participant screening number assigned
* Demographics (including age, gender, ethnicity, number of years in higher education, family history of depression)
* Depression history (as applicable), including age at first episode, number of past episodes of depression and time since last episode
* Brief medical history
* Medication history (current medication, medication taken over the past month, any available information on previous antidepressant medications)
* Entry criteria check Participants that do not meet the entry criteria ('screen failures') will leave the study.

Participants that meet the entry criteria will complete the following activities in the order below:

* Montgomery-Åsberg Depression Rating Scale (MADRS)
* Registration of participant on the Electronic Patient Reported Outcomes(ePRO) system (by study researcher)
* Participant creates ePRO system account
* PReDicT Test (which includes the Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR-16) questionnaire from which baseline QIDS-SR-16 scores are obtained)
* Randomisation (by the ePRO system)
* 5 dimensional - 5 Level quality of life questionnaire (EQ-5D-5L)
* Health Economics Questionnaire (HEQ)
* Oxford CAPabilities questionnaire-Mental Health (OxCAP-MH) (UK and Germany only)
* Social Adjustment Scale - Self-Report (screen version) (SAS-SR (screen version))
* Generalised Anxiety Disorder Questionnaire, 7 item version (GAD-7)
* Digit Symbol Substitution Test (DSST)
* Adverse Events (AEs), Adverse Device Effects (ADEs) and device deficiencies will be recorded from the signing of the ICF and continue until week 8.

At the end of the visit, enrolled participants will be asked to start their prescribed SSRI. Dose and frequency will be as prescribed by their physician.

Visit 2 is only required for participants in the PReDicT arm.

* This visit will take place after PReDicT #2 has been completed. It will preferably take place within 1 day (same day is permissible). The visit may be conducted by telephone (if permitted locally) or at the study site. Visit duration will be approximately 5-10 minutes. The following will take place.
* A study researcher will review the PReDicT Test results online.
* If the PReDicT Test results indicate a positive response to the prescribed antidepressant:

  * Antidepressant treatment is not changed.
  * The next study visit is Visit 4 (there is no Visit 3 for this participant).
* If the PReDicT Test results indicate an insufficient response to the prescribed antidepressant:

  * Antidepressant treatment is altered (by a physician) in accordance with locally appropriate guidelines and judgement of the physician (i.e. normally the dose of the current medication is increased).

Visit 3 is only required for participants in the PReDicT arm who have completed PReDicT #3. This visit will be the same as Visit 2.

Visit 4 (All Participants) The visit will take place 8-10 weeks after starting antidepressant treatment. Visit duration will be approximately 60 minutes. All participants will then continue into the online follow-up phase of the study.

The following Visit 4 activities must be completed at the study site and will take approximately 30 minutes.

* MADRS
* Number and dates of non-study clinical visits for depression since Visit 1
* Review of antidepressant medication compliance. Document all changes to dose or type of antidepressant. Refer to ePRO system data. Ensure any discrepancies between eCRF data and ePRO data are explained
* Review of concomitant medication since last visit
* Review of AEs, ADEs and device deficiencies
* Serious Adverse Events (SAEs) and device-related incidents will be followed up as set out in Section 10.0, Adverse Event Reporting. Non-serious AEs will be followed up at the study physician's discretion The following Visit 4 online questionnaires may be completed at home or at the study site. They can take place before or after the other Visit 4 activities. Questionnaires will take approximately 30 minutes to complete.
* QIDS-SR-16
* EQ-5D-5L
* HEQ
* OxCAP-MH (UK and Germany only)
* SAS-SR (screener version)
* GAD-7
* DSST
* Patient Acceptability Questionnaire An email reminder will be sent to each participant at 8 weeks. An alert will be emailed to the study researcher after 2 days if the questionnaire(s) have not been completed. Researchers should contact the participant as soon as possible and ask them to complete the missing questionnaire(s).

Participants will complete the following online questionnaires every 4 weeks for 40 weeks, starting 4 weeks after Visit 4. The questionnaires take approximately 15 minutes (total) to complete.

* QIDS-SR-16
* EQ-5D-5L
* HEQ Participants will complete the following online questionnaires at week 24 and week 48 of the study.
* OxCAP-MH (UK and Germany only)
* SAS-SR (screener version) For all online questionnaires, an email reminder will be sent to each participant on the day that completion of the questionnaires is due. The email will include a link to the questionnaires on the ePRO system.

An alert will be emailed to the study researchers after 2 days if the questionnaire(s) have not been completed. A researcher will contact the participant as soon as possible and ask them to complete the missing questionnaire(s).

To improve study participation and reduce drop-outs, participants in the PReDicT arm of the study will be able to view their QIDS-SR-16 scores on the ePRO system from Visit 4 up to and including the final online follow-up (Follow-Up #10, occurring 40 weeks after Visit 4).

Prescribing physicians and (if relevant) support staff at each study site will be asked to complete a Healthcare Provider Acceptability Questionnaire at around the time that the final participant at their study site completes Visit 4.

The Healthcare Provider Acceptability Questionnaire is a 40-item questionnaire covering their experience of taking part in the study, their experience of using the PReDicT Test in the study and their future intentions regarding the use of the PReDicT Test. Additional space is provided for free-text comments.

In England and Germany, digitally recorded semi-structured interviews will be performed with maximum variance samples of participants (patients), prescribing physicians and (if relevant) support staff. Interviews will be conducted by fluent speakers of English and/or German (as appropriate) and may be carried out face-to-face or by telephone/Skype.

Interviewees will be selected in such a way that there is appropriate representation of factors including age, gender, questionnaire responses, full- and part-time staff, urban and rural location and high/low/non-recruiting study sites.

Approximately 15 to 20 participants, 20-25 prescribing physicians and a small number of support staff (if relevant) will be interviewed. Interviews will be conducted by trained researchers and will take place during and after completion of the clinical phase of the study, depending on whether participants or study staff are being interviewed. Participants will be recruited for interview within 1 to 2 months after they have completed Visit 4. Prescribing physicians and support staff will be interviewed after the end of the clinical phase at their study site (when all participants have been recruited).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 70 inclusive.
* Diagnosed with a depressive episode by a physician (either first episode or recurrent) and requiring treatment with a selective serotonin reuptake inhibitor (SSRI) medication (excluding fluoxetine).
* Prescribed an SSRI by a physician for the treatment of depression within 7 days prior to Visit 1, but has not yet started taking medication.
* Is intending to start SSRI treatment within 7 days of Visit 1.

Exclusion Criteria:

* Previous history of mania.
* Is currently taking an antidepressant medication or has stopped antidepressant treatment within 2 weeks prior to Visit 1.
* Requires immediate referral to alternative mental health services (e.g. where a patient seen in primary care is referred to secondary care services).
* Presents to a physician with significant current suicidal intent requiring enhanced care.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 913 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Increase in proportion of depressed patients showing a response to treatment at week 8 when using the PReDicT Test to direct antidepressant treatment compared to treatment as usual as measured by the QIDS-SR-16 | 8 weeks
  QIDS-SR-16 is a standard questionnaire "The Quick Inventory of Depressive Symptomatology" (16-Item) (Self-Report). This covers questions on falling asleep, sleep during the night, waking up , sleeping too much, feeling sad ,appetite, weight, concentration , how they view themselves, thoughts of death and suicide, general interests, energy levels, feeling slowed down , feeling restless. These will be compared at baseline and after 8 weeks of treatment.

SECONDARY OUTCOMES:
Compare the change from baseline in QIDS-SR-16 scores | 8 weeks
  To compare the change from baseline in QIDS-SR-16 scores (i.e. treated as a continuous variable) at week 8 between depressed patients receiving treatment directed by the PReDicT Test and those receiving TaU.
Increase in proportion of depressed patients showing a response to treatment at week 8 when using the PReDicT Test to direct antidepressant treatment compared to treatment as usual as measured by a reduction of >50% in the MADRS score | 8 weeks
  • To determine whether use of the PReDicT Test to direct antidepressant treatment results in an increased proportion of depressed patients showing a response to treatment at week 8 compared to TaU, where response is defined as a decrease of 50% or more from baseline MADRS scores.(Montgomery-Åsberg Depression Rating Scale)
Increase in proportion of depressed patients showing remission from depression at week 8 when using the PReDicT Test to direct antidepressant treatment compared to treatment as usual as measured by a QIDS-SR-16 score <=5 | 8 Weeks
  • To determine whether use of the PReDicT Test to direct antidepressant treatment results in an increased proportion of depressed patients achieving remission at week 8 compared to TaU where remission is defined as a QIDS-SR-16 score of 5 or less.
Compare changes in baseline of the QIDS-SR-16 score | 12 weeks
  • To compare the change from baseline in QIDS-SR-16 score (i.e. treated as a continuous variable) at week 12 between depressed patients receiving treatment directed by the PReDicT Test and those receiving TaU.
Compare changes in baseline of the QIDS-SR-16 score | 24 weeks and 48 weeks
  • To compare the change from baseline in QIDS-SR-16 score (i.e. treated as a continuous variable) at 24 and 48 weeks between depressed patients receiving treatment directed by the PReDicT Test and those receiving TaU.
Health economic analysis on societal costs and cost-effectiveness/cost-utility of the PReDicT Test compared with Treatment as Usual as measured by the EQ-5D-5L | 24 weeks and 48 weeks (optional)
  Health economic analysis will include: (i) a detailed patient-level cost analysis of health, social care and other broader societal costs for both the PReDicT and the TaU arms of the study and (ii) an incremental within-trial economic evaluation comparing the PReDicT arm and the TaU arm of the study in terms of their costs and outcomes over the 6 months main trial follow-up period (week 0 to week 24). An optional analysis of the data after 12 months (week 0 to week 48) may also be performed.
Health economic analysis on societal costs and cost-effectiveness/cost-utility of the PReDicT Test compared with Treatment as Usual as measured by the QIDS-SR-16 | 24 weeks and 48 weeks (optional)
  Health economic analysis will include: (i) a detailed patient-level cost analysis of health, social care and other broader societal costs for both the PReDicT and the TaU arms of the study and (ii) an incremental within-trial economic evaluation comparing the PReDicT arm and the TaU arm of the study in terms of their costs and outcomes over the 6 months main trial follow-up period (week 0 to week 24). An optional analysis of the data after 12 months (week 0 to week 48) may also be performed.
Health economic analysis on societal costs and cost-effectiveness/cost-utility of the PReDicT Test compared with Treatment as Usual as measured by the OxCAP-MH | 24 weeks and 48 weeks (optional)
  Health economic analysis will include: (i) a detailed patient-level cost analysis of health, social care and other broader societal costs for both the PReDicT and the TaU arms of the study and (ii) an incremental within-trial economic evaluation comparing the PReDicT arm and the TaU arm of the study in terms of their costs and outcomes over the 6 months main trial follow-up period (week 0 to week 24). An optional analysis of the data after 12 months (week 0 to week 48) may also be performed.
Health economic analysis on societal costs and cost-effectiveness/cost-utility of the PReDicT Test compared with Treatment as Usual as measured by the HEQ | 24 weeks and 48 weeks (optional)
  Health economic analysis will include: (i) a detailed patient-level cost analysis of health, social care and other broader societal costs for both the PReDicT and the TaU arms of the study and (ii) an incremental within-trial economic evaluation comparing the PReDicT arm and the TaU arm of the study in terms of their costs and outcomes over the 6 months main trial follow-up period (week 0 to week 24). An optional analysis of the data after 12 months (week 0 to week 48) may also be performed.
Obtain further feasibility data | 48 weeks
  Acceptability questionnaires will be reported using descriptive statistics. Free text comments will be analysed thematically. Questionnaire and demographic data will be used to guide sampling for the semi-structured interviews.
Assess the acceptability and perceived value of the PReDicT Test | 48 weeks
  Acceptability questionnaires will be reported using descriptive statistics. Free text comments will be analysed thematically. Questionnaire and demographic data will be used to guide sampling for the semi-structured interviews.
Compare the change from baseline in GAD-7 score | 8 Weeks
  To compare the change from baseline in GAD-7 score (i.e. treated as a continuous variable) at week 8 between depressed patients receiving treatment directed by the PReDicT Test and those receiving TaU. (GAD-7: Generalised Anxiety Disorder Questionnaire, 7 item version
Compare the change from baseline on the depression and anxiety items | 8 weeks
  To compare the change from baseline on the depression and anxiety items (analysed separately) of the QIDS-SR-16 at week 8 between depressed patients receiving treatment directed by the PReDicT Test and those receiving TaU by analysis of the QIDS-SR-16 using linear regression to quantify treatment effects with a baseline measure included as a covariate
Determine the change of cognitive function | 8 weeks
  To determine the change of cognitive function (assessed using the DSST) from baseline to week 8 between depressed patients receiving treatment directed by the PReDicT Test and those receiving TaU.
  o DSST: Digit Symbol Substitution Test.
Compare the change from baseline in self-reported social and occupational functioning | weeks 8, 24 and 48
  To compare the change from baseline in self-reported social and occupational functioning at weeks 8, 24 and 48 between depressed patients receiving treatment directed by the PReDicT Test and those receiving TaU.
  * Social and occupational functioning will be assessed by SAS-SR (screener version).
  * SAS-SR: Social Adjustment Scale - Self-Report (screener version). by which will be followed up monthly over the period of one year, multilevel modelling will be conducted to quantify treatment effects with 'participant' as a level two unit, treatment status and treatment x time interactions. Baseline measurement will be included in multilevel model as a covariate
Device safety as required by medical devices legislation | 48 weeks
  Analysis of Safety will be reviewed and reported using descriptive statistics

CONTACTS AND LOCATIONS:
Overall Officials: Mike Browning, Principal Investigator — P1vital Limited
Locations (76):
- Centre Hospitalier Sainte-Anne, Paris, France
- Germany (21):
  - Praxis Dr. Hofmann, Aschaffenburg
  - Praxis Wagner, Aschaffenburg
  - Praxis Dunkel, Frankfurt am Main
  - Agaplesion Markus Krankenhaus, Frankfurt am Main
  - Dept of Psychiatry, Outpatient Clinic, University Hospital, Frankfurt am Main
  - Praxis Dr. Körner, Frankfurt am Main
  - Praxis Dr. Gunreben, Kitzingen
  - Praxis Dr. Boreatti, Lohr
  - Praxis Dr. Vondung, Mühlheim
  - Praxis Bayer, Offenbach
  - Praxis Dr. Frühauf, Offenbach
  - Praxis Schell, Offenbach
  - Praxis Dr. Rost, Randersacker
  - Praxis Dr. Meesmann, Schweinfurt
  - Praxis Habermeyer, Veitshöchheim
  - Schloss Werneck, Werneck
  - Department of Psychiatry, Würzburg
  - Medizinisches Studienzentrum (MSZ), Würzburg
  - Praxis Dr. Heine, Würzburg
  - Praxis Dr. Kropp, Würzburg
  - Praxis Dr. Reimann, Würzburg
- Netherlands (20):
  - Gezondheidscentrum de Keijzer, Amsterdam
  - Gezondheidscentrum Borgerstraat, Amsterdam
  - Gezondheidscentrum De Vaart, Amsterdam
  - GGZ inGeest, Amsterdam
  - Prezens - bGGZ, Amsterdam
  - Gezondheidscentrum Osdorp, Amsterdam
  - Huisartsenpraktijk Houben en Zonneveld, Amsterdam
  - Huisartsenpraktijk Land, Amsterdam
  - Huisartsenpraktijk De Grote Rivieren, Amsterdam
  - Dept of Psychiatry, Vumc, Amsterdam
  - Universitaire Huisartsenpraktijk VUmc, Amsterdam
  - Huisartsenpraktijk MC Gelderlandplein, Amsterdam
  - Huisartsenpraktijk Buitenhof, Amsterdam
  - Gezondheidscentrum Venserpolder, Amsterdam
  - Gezondheidscentrum Klein-Gooioord, Amsterdam
  - Gezondheidscentrum Gein, Amsterdam
  - Gezondheidscentrum Reigersbos, Amsterdam
  - Gezondheidscentrum Nellestein, Amsterdam
  - Gezondheidscentrum Diemen-Noord, Amsterdam
  - De Hoofdlijn, IJmuiden
- Spain (5):
  - CAP Barceloneta, Barcelona
  - Hospital del Mar, Barcelona
  - CAP Vila Olímpica, Barcelona
  - Centre Fòrum, Barcelona
  - CAP Larrard, Barcelona
- United Kingdom (29):
  - St Chad's Surgery, Midsomer Norton, Bath
  - The Boathouse Surgery, Pangbourne, Berkshire
  - Carlisle Healthcare, Carlisle, Cumbria
  - The Limes Medical Centre, Alfreton, Derbyshire
  - Burbage Surgery, Burbage, Leicestershire
  - Lindum Medical Practice, Lincoln, Lincolnshire
  - Nettleham Medical Practice, Nettleham, Lincoln
  - Welton Family Health Centre, Welton, Lincoln
  - Lakeside Surgery, Corby, Northamptonshire
  - Danetre Medical Practice, Daventry, Northamptonshire
  - Earls Barton Medical Centre, Earls Barton, Northamptonshire
  - Rothwell and Desborough Healthcare Group, Rothwell, Northamptonshire
  - Albany House Medical Centre, Wellingborough, Northamptonshire
  - Atherstone Surgery, Atherstone, Warwickshire
  - Sherbourne Medical Centre, Royal Leamington Spa, Warwickshire
  - The Porch Surgery, Corsham, Wiltshire
  - Adcroft Surgery, Trowbridge, Wiltshire
  - Bradford Road Medical Centre, Trowbridge, Wiltshire
  - Westbury Group Medical Practice, Westbury, Wiltshire
  - The Pulteney Practice, Bath
  - Newton Place Surgery, Faversham
  - Thurmaston Health Centre, Leicester
  - Birchwood Medical Practice, Lincoln
  - Lincoln University Health Care, Lincoln
  - Leicester Terrace, Northampton
  - Danes Camp Practice, Northampton
  - Family Medical Centre, Nottingham
  - University of Nottingham Health Service - Cripps Health Centre, Nottingham
  - South Oxford Health Centre, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] World Health Organization, The Global Burden of Disease: 2004 update. nDeneva, World Health Organization, 2008.
- [Result] Wittchen HU, Jacobi F, Rehm J, Gustavsson A, Svensson M, Jonsson B, Olesen J, Allgulander C, Alonso J, Faravelli C, Fratiglioni L, Jennum P, Lieb R, Maercker A, van Os J, Preisig M, Salvador-Carulla L, Simon R, Steinhausen HC. The size and burden of mental disorders and other disorders of the brain in Europe 2010. Eur Neuropsychopharmacol. 2011 Sep;21(9):655-79. doi: 10.1016/j.euroneuro.2011.07.018. PMID 21896369
- [Result] Rush AJ. STAR*D: what have we learned? Am J Psychiatry. 2007 Feb;164(2):201-4. doi: 10.1176/ajp.2007.164.2.201. No abstract available. PMID 17267779
- [Derived] Kingslake J, Dias R, Dawson GR, Simon J, Goodwin GM, Harmer CJ, Morriss R, Brown S, Guo B, Dourish CT, Ruhe HG, Lever AG, Veltman DJ, van Schaik A, Deckert J, Reif A, Stablein M, Menke A, Gorwood P, Voegeli G, Perez V, Browning M. The effects of using the PReDicT Test to guide the antidepressant treatment of depressed patients: study protocol for a randomised controlled trial. Trials. 2017 Nov 23;18(1):558. doi: 10.1186/s13063-017-2247-2. PMID 29169399